CLINICAL TRIAL: NCT03983603
Title: Plant Stanol Esters in the Prevention of Clinical Symptoms Related to Asthma: The PLANTASTIC Trial
Brief Title: Plant Stanol Esters and Preventing Asthma Symptoms
Acronym: PLANTASTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Raisio Group (Industry); TKI Life Sciences and Health (LSH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 18-064
Record Dates: First submitted 2019-06-04; First posted 2019-06-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-02

CONDITIONS: Asthma, Allergic; Cardiovascular Diseases
Keywords: Plant stanols; Asthma; Immune system; Metabolic health
MeSH Terms: conditions — Asthma; Cardiovascular Diseases | interventions — Parturition; plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant stanol group (Experimental): This arm receives soft chews containing 0.5g of plant stanols (delivered as plant stanol esters).
  Interventions: Dietary Supplement: Soft chews containing 0.5g plant stanols (delivered as plant stanol esters)
- Placebo group (Placebo Comparator): This arm receives soft chews that do not contain 0.5g of plant stanols (delivered as plant stanol esters).
  Interventions: Dietary Supplement: Placebo soft chew

INTERVENTIONS:
Dietary Supplement: Soft chews containing 0.5g plant stanols (delivered as plant stanol esters) — Soft chews containing 0.5g plant stanols delivered as plant stanol esters
  Arms: Plant stanol group
Dietary Supplement: Placebo soft chew — Soft chew that does not contain plant stanols
  Arms: Placebo group

SUMMARY:
Plant stanols are known to lower low-density lipoprotein cholesterol. However, studies have suggested that these compounds also influence the immune system. Asthmatic responses are predominantly T helper (Th)2 cell dependent, while plant stanols were previously found to activate Th1 cells and shift the immune response away from the Th2 cell dominant asthmatic response. The question now is whether this also translates into a reduction of clinical symptoms in asthma patients.The primary objective of this study is to demonstrate clinical benefits of prolonged consumption of plant stanols (delivered via plant stanol esters) in asthma patients. The secondary objectives are to evaluate the mechanisms via which plant stanols modulate the immune system and to evaluate the effects of plant stanol ester consumption on cardiovascular (CVD) risk parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with allergic asthma (GINA step 1-4) which is in a stable phase at the moment of inclusion (defined as no changes in asthma control and lung function in (at least) the past three months)
* Have been treated with prescribed asthma medication for at least one year
* Aged 18-70 years old
* BMI between 20 and 35 kg/m2
* Willing to abstain from products containing plant sterols or stanols one month prior to the study (products with a cholesterol lowering claim of Becel ProActiv, Benecol, Danacol, store brands)
* Willing to abstain from products containing plant sterols or stanols during the study (products with a cholesterol lowering claim of Becel ProActiv, Benecol, Danacol, store brands)
* Willing to keep the intake of fish oil supplements constant

Exclusion Criteria:

* Currently smoking or quitted smoking in the past year, with a maximum of 10 packyears as smoking history (packyears = packs per day * years of smoking)
* Allergy to an ingredient of the soft chews
* Suffering from inflammatory diseases (for CVD, illness must be minimally 3 years ago and currently under control in order to participate in the study)
* Fasting plasma glucose > 7.0 mmol/L
* Fasting serum TC > 8.0 mmol/L
* Having donated blood within one month prior to the start of the study, or planning to donate blood during the study
* Pregnant women
* Breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Asthma control questionnaire score | Change between T=0 months and T=12 months
  The ACQ consists of seven questions: five questions are on asthma related symptoms, one on medication use and one on the FEV1. Participants are asked to score their symptoms and medication use of the past week on a scale from zero to six. The score of the ACQ is the average score on the seven questions. A score of zero means that asthma is fully controlled; a score of six means that asthma is severely uncontrolled. The minimal clinically important difference is 0.5. The ACQ has been validated and is widely use in research and clinical settings.

SECONDARY OUTCOMES:
Asthma control questionnaire score | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  The ACQ consists of seven questions: five questions are on asthma related symptoms, one on medication use and one on the FEV1. Participants are asked to score their symptoms and medication use of the past week on a scale from zero to six. The score of the ACQ is the average score on the seven questions. A score of zero means that asthma is fully controlled; a score of six means that asthma is severely uncontrolled. The minimal clinically important difference is 0.5. The ACQ has been validated and is widely use in research and clinical settings.
Forced expiratory volume in 1 second | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Amount of air that can be exhaled forcefully in one second in Liters or %
Forced vital capacity | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Amount of air that can be exhaled forcefully in total in Liters or %
Asthma related medication use | Throughout 1 year
  Self-reported medication use
Number of visits to the general practitioner or hospital | Throughout 1 year
  Self-reported amount of visits to the general practitioner or hospital
Incidence counts of exacerbations and other asthma related complaints | Throughout 1 year
  Self-reported amount of exacerbations and other asthma related complaints
Duration of exacerbations | Throughout 1 year
  Self-reported duration of exacerbations
Severity of exacerbations | Throughout 1 year
  Self-reported severity of exacerbations
Calculated disease load | Throughout 1 year
  Number x duration of exacerbations
Number of infections that occur throughout the study | Throughout 1 year
  Self-reported amount of infections
Leukocyte count | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Number of leukocytes measured in EDTA plasma
Leukocyte differential count | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Number of subgroups of leukocytes measured in EDTA plasma
Red blood cell count | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Number of red blood cells measured in EDTA plasma
Platelet count | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Number of platelets measured in EDTA plasma
Hematocrit | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Hematocrit measured in EDTA plasma
Hemoglobin | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Hemoglobin measured in EDTA plasma
Immune parameters (1) | T=0 months, T=6 months, T=12 months
  Cytokine production by PBMCs after stimulation with antiCD3-antiCD28 antiCD28 antibodies using the TruCulture system
Immune parameters (2) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Total IgE
Immune parameters (3) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Total IgM
Immune parameters (4) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  hsCRP
Fasted metabolism (1) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Serum lipid and lipoprotein profile
Fasted metabolism (2) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Serum non-cholesterol sterols and stanols
Fasted metabolism (3) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Plasma glucose metabolism
Vascular function markers (1) | T=0 months and T=12 months
  Carotid-femoral pulse wave velocity (PWV)
Vascular function markers (2) | T=0 months and T=12 months
  Pulse wave analysis (PWA)
Vascular function markers (3) | T=0 months and T=12 months
  Retinal microvascular caliber
Cardiometabolic risk marker | T=0 months and T=12 months
  Office blood pressure
Cognitive function | T=0 months and T=12 months
  CANTAB tests
Anthropometry (1) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Body weight
Anthropometry (2) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Height
Anthropometry (3) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Body mass index
Anthropometry (4) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Waist circumference
Anthropometry (5) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Hip circumference
Anthropometry (6) | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Waist-to-hip ratio
Quality of life score | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  32-item questionnaire (including social, spiritual, emotional, cognitive, physical, activities of daily living, and integrated Quality of Life)
Fatigue | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Fatigue severity score (FSS), a 9-item questionnaire is used to determine the severity of fatigue a subject experienced in the past week during daily activities
Physical activity | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Baecke's questionnaire
Mood | T=0 months, T=3 months, T=6 months, T=9 months, T=12 months
  Affect grid
Diet | T=0 months, T=6 months, T=12 months
  Food frequency questionnaire is used to determine if the participants maintain their habitual diet and to determine if the participants do not consume plant stanols and/or sterols outside the intervention
Immune cell characterisation | T=0 months, T=6 months, T=12 months
  Fluorescence-activated cell sorting (FACS)

OTHER OUTCOMES:
Mechanistic outcomes for measuring the immune response | Weekly from T=12 months to T=13 months
  Vaccination response to vaccines against tetanus, pneumococcal bacteria and rabies

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, PhD, Principal Investigator — Maastricht University Medical Center; Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands